CLINICAL TRIAL: NCT03276130
Title: Management of Health-Related Quality of LIfe Impairment, Including Pain, Depression and Anxiety, in People With Haemophilia A and B
Brief Title: Management of Health-Related QoL Impairment, Including Pain, Depression and Anxiety, in People With Haemophilia A and B
Acronym: MIND
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.HAEM89-003
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Haemophilia A; Haemophilia B
Keywords: Blood coagulation disorder; Haematologic diseases; Coagulation protein disorder; Hemorrhagic disorder; Genetic diseases, inborn; Pain; Anxiety; Pain medication; Anxiety medication
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Blood Coagulation Disorders; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Part A: Retrospective register study: To describe the usage of prescribed pain, anti-depressive and anti-anxiety medication during a 10-year period based on retrospective data from patient and drug registries. Population: All People with Haemophilia A and B identified through national administrative register or from local register at each treatment centre. The People with Haemophilia group will be compared against an age and gender matched control group from the general population.
- Part B1: Survey to HTC: The survey will be sent out to the relevant physician at each Haemophilia Treatment Centers (HTC) with direct and frequent patient contacts.
- Part B2: Survey to PwH: All People with Haemophilia (PwH) listed at HTCs will be invited to participate in the patient survey.

SUMMARY:
The puropse of this non-interventional register and survey study is to identify the patterns of prescribed pain, anti-depressive and anti-anxiety medication and management of pain, depression and anxiety for people with haemophilia. The study will be conducted in the Nordic countries (Sweden, Norway, Denmark, Finland) and the aim is to cover the entire haemophilia population in the register part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Part A population will be defined by having:
* at least one health care contact with main diagnosis haemophilia A or haemophilia B, and/or;
* at least one prescription of factor VIII or factor IX concentrates, or;
* bypassing agents used in the treatment of PwH during the inclusion period.
* Part B1 population: Relevant physician at each HTC with direct and frequent patient contact.
* Part B2 population: PwH 5 years or older listed at participating HTCs

Exclusion Criteria:

* NA

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All PwH in Sweden, Norway, Denmark and Finland
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Use of medication for pain, depression and anxiety (yes/no?) | Retrospectively 10 years
  Based on Registry data
Annualised consumption of pain medications as assessed by filled prescription | Retrospectively 10 years
  Based on Registry data
Annualised consumption of anti-anxiety medications as assessed by filled prescription | Retrospectively 10 years
  Based on Registry data
Annualised consumption of anti-depressive medications as assessed by filled prescription | Retrospectively 10 years
  Based on Registry data
Duration of pain medications as measured by expected doses of medicines. | Retrospectively 10 years
  Based on Registry data
Duration of anti-depressive medications as measured by expected doses of medicines. | Retrospectively 10 years
  Based on Registry data
Duration of anti-anxiety medications as measured by expected doses of medicines. | Retrospectively 10 years
  Based on Registry data
Pharmacological and non-pharmacological treatments for management of Health-Related Quality of Life (HRQoL) impairment, including treatment of pain | Inclusion in survey study
  Assessed by Health Care Professional (HCP) survey in Part B1
Pharmacological and non-pharmacological treatments for management of HRQoL impairment, including treatment of anxiety | Inclusion in survey study
  Assessed by HCP survey in Part B1
Pharmacological and non-pharmacological treatments for management of HRQoL impairment, including treatment of depression | Inclusion in survey study
  Assessed by HCP survey in Part B1
The perspective and experience of HCPs with direct and frequent patient Contacts on the strategies for the management of HRQoL impairment, including treatment of pain at each Haemophlia Treatment Centre | Inclusion in survey study
  Assessed by HCP survey in Part B1
The perspective and experience of HCPs with direct and frequent patient Contacts on the strategies for the management of HRQoL impairment, including treatment of anxiety at each Haemophlia Treatment Centre | Inclusion in survey study
  Assessed by HCP survey in Part B1
The perspective and experience of HCPs with direct and frequent patient Contacts on the strategies for the management of HRQoL impairment, including treatment of depression at each Haemophlia Treatment Centre | Inclusion in survey study
  Assessed by HCP survey in Part B1
Self-reported current and previous use of medications for pain | Inclusion in survey study
  Assessed by patient survey in Part B2
Self-reported current and previous use of medications for anxiety | Inclusion in survey study
  Assessed by patient survey in Part B2
Self-reported current and previous use of medications for depression | Inclusion in survey study
  Assessed by patient survey in Part B2
Social and physical activity level | Inclusion in survey study
  Assessed by patient survey in Part B2
Euro-QoL 5 Dimensions 5 Levels (EQ-5D-5L) | Inclusion in survey study
  Assessed by patient survey in Part B2
Patient satisfaction with current management of pain | Inclusion in survey study
  Assessed by patient survey in Part B2
Patient satisfaction with current management anxiety | Inclusion in survey study
  Assessed by patient survey in Part B2
Patient satisfaction with current management of depression | Inclusion in survey study
  Assessed by patient survey in Part B2
Patient satisfaction of received treatment for pain | Inclusion in Survey study
  Assessed by patient survey in Part B2
Patient satisfaction of received treatment for anxiety | Inclusion in Survey study
  Assessed by patient survey in Part B2
Patient satisfaction of received treatment for depression | Inclusion in Survey study
  Assessed by patient survey in Part B2

CONTACTS AND LOCATIONS:
Locations (5):
- Swedish Orphan Biovitrum Research Site, Copenhagen, Denmark
- Swedish Orphan Biovitrum Research Site, Helsinki, Finland
- Sweden (3):
  - Swedish Orphan Biovitrum Research Site, Gothenburg
  - Swedish Orphan Biovitrum Research Site, Malmo
  - Swedish Orphan Biovitrum Research Site, Stockholm

REFERENCES:
- [Derived] Steen Carlsson K, Astermark J, Baghaei F, Brodin E, Funding E, Holmstrom M, Osterholm K, Bergenstrale S, Lethagen S. Comorbidity and Mortality in Men and Women With Haemophilia in Three Nordic Countries-Comparisons to Matched Controls. Haemophilia. 2025 May;31(3):401-411. doi: 10.1111/hae.70023. Epub 2025 Mar 18. PMID 40099856
- [Derived] Steen Carlsson K, Winding B, Astermark J, Baghaei F, Brodin E, Funding E, Holmstrom M, Osterholm K, Bergenstrale S, Andersson E, Lethagen S. Pain, depression and anxiety in people with haemophilia from three Nordic countries: Cross-sectional survey data from the MIND study. Haemophilia. 2022 Jul;28(4):557-567. doi: 10.1111/hae.14571. Epub 2022 Apr 23. PMID 35460313